CLINICAL TRIAL: NCT06357208
Title: IMPACT OF BREATH CONTROL AND RETENTION ON PATIENT STRESS. E.S IN MEDICALLY ASSISTED REPRODUCTION BREATH HOLD TO BREATH BETTER PROGRAM IN MEDICALLY ASSISTED REPRODUCTION
Brief Title: IMPACT OF BREATH CONTROL AND RETENTION ON PATIENT STRESS. E.S IN MEDICALLY ASSISTED REPRODUCTION
Acronym: BHBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-AOI-06; 2023-A02687-38 (Other: ANSM)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Reproductive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Control and Retention (Experimental): Breathing Control and Retention
  Interventions: Other: Breathing Control and Retention
- Usual follow-up (No Intervention): the patient come at the begin of the study and come back after one month

INTERVENTIONS:
Other: Breathing Control and Retention — 4 appointments with training of Breathing Control and Retention
  Other Names: respiratory exercice
  Arms: Breathing Control and Retention

SUMMARY:
the investigator propose for patient in the course of Medically Assisted Reproduction a study with to arm: one arm active "Breathing Control and Retention" and the other arm control

DETAILED DESCRIPTION:
After signing the informed consent, the patient makes an appointment for an exchange with the psychologist at the Reproduction center.

During this exchange, the psychologist gives him the evaluation scales, explains to him when to complete them and re-explains the progress of the study.

Patients in the active "Breathing Control and Retention" group make 4 appointments, one week apart, with the Bluenery Academy. The participants self-assess 2 days before starting the breathing program (M0), 2 days after the end of the program, 1 month after starting the program (M1).

Patients in the "Usual follow-up" control group complete the self-assessments 2 days after the discussion with the psychologist (M0) and 1 month later (M1).

At the end of the 2 assessments, the patient was included. sends his assessment book to the psychologist.

An appointment will be made after the rating to communicate the results to them.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried woman and couple of women with societal infertility,
* couple with medical infertility defined as absence of pregnancy after 12 months without contraception,
* age greater than 18 years,
* patient who has signed informed consent and affiliated to social security.
* Patient available at the proposed slots over 4 weeks

Exclusion Criteria:

* pregnant women before starting the program,
* heart failure
* Thrombocytopenia
* epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of stressed patients | month 1
  with score of 27 on the Perceived Stress Scale

SECONDARY OUTCOMES:
STAI Y-A (anxiety state) scale | month 1
  feeling anxious at the time with a score > 39 for men and > 47 for women

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BENOIT, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No